CLINICAL TRIAL: NCT01128478
Title: Early Enteral Tube Feeding Compared With Pancreas Rest in Patients With Acute Pancreatitis: a Randomized Controlled Trial
Brief Title: MIld to MOderate Acute Pancreatitis: Early naSogastric Tube Feeding Compared With pAncreas Rest (MIMOSA)
Acronym: MIMOSA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Max Petrov, Principal Investigator, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NTX/08/11/107
Record Dates: First submitted 2010-05-11; First posted 2010-05-24 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Acute Pancreatitis
Keywords: Acute pancreatitis; Enteral nutrition; Pancreas rest
MeSH Terms: conditions — Pancreatitis | interventions — Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enteral tube feeding (Other): Nasogastric tube feeding started within 24 h of hospital admission
  Interventions: Procedure: Enteral tube feeding
- Nil-per-mouth regimen (No Intervention): Conventional management

INTERVENTIONS:
Procedure: Enteral tube feeding — Nasogastric tube feeding started within 24 h of hospital admission
  Arms: Enteral tube feeding

SUMMARY:
Pain relapse during oral refeeding occurs in at least one-fifth of patients with acute pancreatitis. The study hypothesis is that early administered enteral tube feeding might reduce a risk of pain relapse and shorten the length of hospital stay in patients with acute pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of acute pancreatitis
* age 18 years or older
* written informed consent

Exclusion Criteria:

* > 96 hours after onset of symptoms
* > 24 hours after hospital admission
* organ failure by the time of randomization
* infectious complications before randomization
* received artificial nutrition before randomization
* previously enrolled into the trial
* chronic pancreatitis
* post-ERCP pancreatitis
* intraoperative diagnosis of acute pancreatitis
* pregnancy
* malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-05; Primary Completion 2011-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | Up to 3 months

SECONDARY OUTCOMES:
Pain relapse | Up to 3 months
Local and systemic complications | Up to 3 months
Feeding intolerance | Up to 3 months
Time to solid oral food tolerated | Approx. one week
Pain-free time | Up to 3 months
Hospital readmission | Up to 6 months
Quality of life | Up to 6 months
Mortality | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Max Petrov, MD, MPH (Epi), Principal Investigator — Universioty of Auckland
Locations (1):
- University of Auckland, Auckland, New Zealand

REFERENCES:
- [Background] Petrov MS. Enteral nutrition: goody or good-for-nothing in acute pancreatitis? Am J Gastroenterol. 2007 Aug;102(8):1828-9; author reply 1829-30. doi: 10.1111/j.1572-0241.2007.01361.x. No abstract available. PMID 17686077
- [Background] Petrov MS, van Santvoort HC, Besselink MG, Cirkel GA, Brink MA, Gooszen HG. Oral refeeding after onset of acute pancreatitis: a review of literature. Am J Gastroenterol. 2007 Sep;102(9):2079-84; quiz 2085. doi: 10.1111/j.1572-0241.2007.01357.x. Epub 2007 Jun 16. PMID 17573797
- [Background] Petrov MS. To feed or not to feed early in acute pancreatitis: still depend on severity? Clin Nutr. 2008 Apr;27(2):317-8. doi: 10.1016/j.clnu.2008.01.011. Epub 2008 Mar 10. No abstract available. PMID 18331767
- [Derived] Petrov MS, McIlroy K, Grayson L, Phillips AR, Windsor JA. Early nasogastric tube feeding versus nil per os in mild to moderate acute pancreatitis: a randomized controlled trial. Clin Nutr. 2013 Oct;32(5):697-703. doi: 10.1016/j.clnu.2012.12.011. Epub 2012 Dec 31. PMID 23340042